CLINICAL TRIAL: NCT02405611
Title: A Multi-component Intervention on Improving Fruit and Vegetable Consumption in Teenagers and Their Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Assistant Professor, Department of Public Health, Qazvin University of Medical Sciences, Qazvin, Iran., Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 682
Record Dates: First submitted 2015-03-25; First posted 2015-04-01 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Nutrition

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- active control (Active Comparator): mothers and children are in active control group and only receive the questionnaires
  Interventions: Behavioral: primary eduction
- mother and student (Experimental): an intervention group in which mothers and children receive the intervention and questionnaires
  Interventions: Behavioral: behavioral
- children (Experimental): only the children receive the intervention and mothers and children receive the questionnaires
  Interventions: Behavioral: behavioral

INTERVENTIONS:
Behavioral: behavioral — The intervention package contains behavior change techniques targeting outcome expectancy, self-efficacy, action planning, coping planning, and self-monitoring. The active control group receives an information sheet regarding recommendations on fruit and vegetable intake. There will be 3 assessment points in time, with 1 month and six months in between. All the intervention materials and information sheets will be handed to participants after the baseline assessment. The self-monitoring calendar will be collected at time 2 assessment.
  Arms: mother and student
Behavioral: behavioral — The intervention package contains behavior change techniques targeting outcome expectancy, self-efficacy, action planning, coping planning, and self-monitoring. The active control group receives an information sheet regarding recommendations on fruit and vegetable intake. There will be 3 assessment points in time, with 1 month and six months in between. All the intervention materials and information sheets will be handed to participants after the baseline assessment. The self-monitoring calendar will be collected at time 2 assessment.
  Arms: children
Behavioral: primary eduction — The intervention package contains behavior change techniques targeting outcome expectancy, self-efficacy, action planning, coping planning, and self-monitoring. The active control group receives an information sheet regarding recommendations on fruit and vegetable intake. There will be 3 assessment points in time, with 1 1 month and six months in between. All the intervention materials and information sheets will be handed to participants after the baseline assessment. The self-monitoring calendar will be collected at time 2 assessment.
  Arms: active control

SUMMARY:
This study is a longitudinal controlled trial that is designed to investigate the effectiveness of a multi-component intervention on improving fruit and vegetable consumption in teenagers and their mothers.

DETAILED DESCRIPTION:
This study is a longitudinal controlled trial that is designed to investigate the effectiveness of a multi-component intervention on improving fruit and vegetable consumption in teenagers and their mothers. Participants will be allocated in three groups with a) an intervention group in which mothers and children receive the intervention and questionnaires, b) only the children receive the intervention and mothers and children receive the questionnaires, and c) mothers and children are in active control group and only receive the questionnaires. The intervention package contains behavior change techniques targeting outcome expectancy, self-efficacy, action planning, coping planning, and self-monitoring. The active control group receives an information sheet regarding recommendations on fruit and vegetable intake. There will be 3 assessment points in time, with 1 months in between. All the intervention materials and information sheets will be handed to participants after the baseline assessment. The self-monitoring calendar will be collected at time 2 assessment.

The primary outcome of this study is to estimate the dyadic mechanisms between mothers and their children regarding improving fruit and vegetable intake. Secondary outcome is to investigate whether fruit and vegetable consumption did improve in the intervention groups in general and also to find the psychological mechanism behind the changes during the time of the study.

ELIGIBILITY:
Inclusion Criteria:

* They are not involved in the nutritional education
* Ability to understand Persian language Adolescents attending high schools in Qazvin

Exclusion Criteria:

* Does not meet inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
changes in fruit intake using a self-reported questionnaire | baseline, 1 Months, 6 months follow-up
  using a self-reported questionnaire
changes in vegetable intake using a self-reported questionnaire | baseline, 1 Months, 6 months follow-up
  using a self-reported questionnaire

SECONDARY OUTCOMES:
changes in self efficacy using a self-reported questionnaire | baseline, 1 Months, 6 months follow-up
  using a self-reported questionnaire
changes in outcome expectancy using a self-reported questionnaire | baseline, 1 Months, 6 months follow-up
  using a self-reported questionnaire
changes in coping planning using a self-reported questionnaire | baseline, 1 Months, 6 months follow-up
  using a self-reported questionnaire
changes in action planning using a self-reported questionnaire | baseline, 1 Months, 6 months follow-up
  using a self-reported questionnaire
changes in self-monitoring using a self-reported questionnaire | baseline, 1 Months, 6 months follow-up
  using a self-reported questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Department of Public Health, Qazvin University of Medical Sciences, Qazvin, Qazvin Province
  - The Organization for Education, Qazvin, Qazvin Province